CLINICAL TRIAL: NCT02662829
Title: Preventing Childhood Tuberculosis in Lesotho (PREVENT Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAN7358; K01AI104351 (NIH)
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Tuberculosis
Keywords: Lesotho; tuberculosis; TB; HIV; adherence; community-based intervention; retention
MeSH Terms: conditions — Tuberculosis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community-based intervention (CBI) (Experimental): 1. Nurse training and mentorship in TB prevention using clinical algorithm based on national guidelines.
  2. Health education using a treatment literacy curriculum for parents and guardians.
  3. Community outreach by trained village health workers.
  Interventions: Behavioral: Community-based intervention
- Standard of Care (SOC) (Active Comparator): At SOC clinics, patients will receive usual care for management of contact tracing, screening, and IPT provision. Childhood TB in Lesotho is managed by nurses in health centers. Per national guidelines, TB patients are asked to bring in child contacts, who are screened using a simple symptom questionnaire. Children who screen negative are assessed for IPT eligibility. Absent contra-indications (eg, active hepatitis, regular alcohol consumption, peripheral neuropathy), nurses counsel children and guardians on IPT benefits, potential side effects, and importance of adherence. Children requiring chest x-rays or gastric lavage and HIV-infected children under age 1 are referred to the hospital. After initiation, patients and guardians return to the clinic monthly for monitoring for side effects, TB symptoms, adherence, and 30-day supply of isoniazid. If adherence problems are noted, the nurse counsels patient and guardian as appropriate.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: Community-based intervention
  Other Names: CBI
  Arms: Community-based intervention (CBI)
Other: Standard of care
  Other Names: SOC
  Arms: Standard of Care (SOC)

SUMMARY:
Lesotho, a small, landlocked country completely surrounded by South Africa, is among the world's poorest nations with one of the world's most severe epidemics of tuberculosis (TB) and HIV. TB incidence is the world's highest and approximately 76% of TB patients are HIV coinfected. Data from similar settings suggest that TB incidence in children is approximately 50% of adult TB incidence. The Lesotho National TB Program has adopted World Health Organization's (WHO) isoniazid preventive therapy (IPT) recommendations for child contacts; however, as in other countries in the region, implementation of IPT in children is limited, no clear strategies guide child contact tracing and screening, and no clear methods ensure provision of IPT in children. Thus, it is important to evaluate novel methods to prevent TB in child contacts of adult TB cases.

The purpose of the PREVENT Study is to identify an effective and acceptable intervention that addresses programmatic, structural and psychosocial barriers to contact tracing, screening, and IPT for child contacts of TB patients, with the ultimate goal of improving health outcomes among children in Lesotho. The study is a two-arm cluster randomized trial, randomized at the TB clinic level, which includes ten TB clinics in Berea district. Clinics are randomized to deliver the community-based intervention (CBI) or standard of care (SOC), with stratification by facility type. The experimental intervention will be delivered to all child contacts of adult TB patients in TB clinics randomly assigned to CBI. In TB clinics assigned to SOC, usual care procedures for contact tracing and IPT will be delivered.

DETAILED DESCRIPTION:
The study intervention, community-based intervention (CBI), will contain multiple components, including: 1) Facility Providers. Providers will be trained on study interventions; job aids will be provided. Nurses will use a clinical algorithm based on national guidelines for intensive case finding and screening of child contacts for TB to assess patients without TB symptoms for IPT eligibility; to initiate IPT; and to monitor for side effects, TB symptoms, and adherence. If a child contact develops TB symptoms during IPT, national guidelines will be followed. HIV testing will be strongly promoted in child contacts. Use of simple available clinic IPT registers will be promoted. The PI will establish systems to track IPT use at monthly multi-disciplinary team meetings; clinic staff will review IPT monitoring data for prior months, identify challenges, and develop solutions. IPT registers will link IPT outcome data to TB register data for index cases. 2) Patients and Guardians. Nurses will explain to patients and guardians that IPT can prevent TB, promote IPT initiation, assess IPT adherence and side effects, and encourage follow-up with village health workers (VHW). Nurses will emphasize HIV testing for children. The VHW role will encompass social support, system navigation, referrals, and advocacy. VHW will follow up with guardians of children who miss appointments or report nonadherence, using scripted, illustrated flipcharts targeting children and guardians. VHW will emphasize to guardians the importance of IPT, encourage IPT and visit adherence, offer support and empathy, provide referrals, and advocate for patients. 3) Community Outreach. To investigate household contacts, VHW will visit homes of all adult TB cases at facilities assigned to CBI. All HIV-infected children and children under 5, regardless of HIV status, will be referred to health facilities. VHW will administer TB symptom screening in child contacts in the community, accompany them and their guardians to the clinic, and provide education sessions, support groups, and adherence counseling.

Study assessments include: 1) outcome data via medical records; 2) pre- and post-intervention interviews with providers; 3) post-intervention guardian interviews; and 4) program characteristics data. Stakeholders and policy makers will be engaged early in the process to help ensure successful integration of findings in programmatic contexts. A dissemination strategy will be developed in consultation with stakeholders and will help ensure scaling up of the intervention, if found effective.

All clinical care, including implementation of the combination intervention package at sites randomized to CIP, will be performed by Lesotho Ministry of Health clinic staff (nurses and VHW). All study procedures, including participant interviews, medical record abstraction, and program characteristics surveys will be performed by study staff.

ELIGIBILITY:
The randomized trial will include review of medical records of all adult TB cases who start TB treatment during the study period.

Providers inclusion criteria:

1. Nurse or village healthcare worker(VHW) working in a CBI clinic or VHW working in the community and affiliated with CBI clinic
2. Aged 18 or older
3. English- or Sesotho speaking
4. Capable of informed consent

Guardians inclusion criteria:

1. Guardian of a child contact
2. Aged 18 or older
3. English- or Sesotho speaking
4. Capable of informed consent

Two groups of guardians will be enrolled: guardians who brought their children for TB screening, and guardians who did not bring their children for TB screening.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2015-12; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Yield of child contacts | 3 years
  Number of child contacts per pulmonary TB case screened, based on review of clinic registers
Percentage of IPT initiation | 3 years
  Percentage of child contacts identified through contact tracing of new adult TB cases during observation period who initiate IPT, based on review of clinic registers
Percentage of IPT completion | Up to 9 months after IPT initiation
  Percentage of child contacts who complete IPT of those who initiate as determined by provider and recorded in clinic charts

SECONDARY OUTCOMES:
Percentage of HIV testing | 3 years
  Percentage of child contacts identified through contact tracing of new adult TB cases during observation period who are tested for HIV, based on review of clinic registers

CONTACTS AND LOCATIONS:
Overall Officials: Yael Hirsch-Moverman, PhD, Principal Investigator — Columbia University
Locations (10):
- Lesotho (10):
  - Berea Hospital, Berea, Berea
  - Holy Family Health Center, Berea, Berea
  - Khubetsoana Health Center, Berea, Berea
  - Koali Health Center, Berea, Berea
  - Kolojane Health Center, Berea, Berea
  - Maluti Hospital, Berea, Berea
  - Pilot Health Center, Berea, Berea
  - St Magdalena Health Center, Berea, Berea
  - St. David Health Center, Berea, Berea
  - St. Theresa Health Center, Berea, Berea

REFERENCES:
- [Derived] Hirsch-Moverman Y, Howard AA, Frederix K, Lebelo L, Hesseling A, Nachman S, Mantell JE, Lekhela T, Maama LB, El-Sadr WM. The PREVENT study to evaluate the effectiveness and acceptability of a community-based intervention to prevent childhood tuberculosis in Lesotho: study protocol for a cluster randomized controlled trial. Trials. 2017 Nov 21;18(1):552. doi: 10.1186/s13063-017-2184-0. PMID 29157275